CLINICAL TRIAL: NCT05960773
Title: Phase II Evaluation of Decitabine/Cedazuridine (INQOVI), an Oral DNA Demethylating Agent in Subjects With BAP1 Cancer Predisposition Syndrome and Subclinical, Early-Stage Mesothelioma
Brief Title: Decitabine/Cedazuridine (INQOVI), an Oral DNA Demethylating Agent, in Subjects With BAP1 Cancer Predisposition Syndrome and Subclinical, Early-Stage Mesothelioma
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: On hold pending updates to the drug/manufacturer information.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10001549; 001549-C
Record Dates: First submitted 2023-07-22; First posted 2023-07-27 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12-19

CONDITIONS: Mesothelioma; Malignant Mesothelioma (MM); Early-stage Mesothelioma; Subclinical Mesothelioma; BRCA1-Associated Protein-1 (BAP1) Mutations; Early-stage BAP1-associated Malignancies
Keywords: BRCA1-Associated Protein-1; CPDS; DNA methyltransferases (DNMT); DNMT1; ring finger domains 1 (UHRF1); germline antigens; peripheral immune subsets
MeSH Terms: conditions — Mesothelioma; Mesothelioma, Malignant | interventions — decitabine and cedazuridine drug combination

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1/ Arm 1 (Experimental): Decitabine/cedazuridine (35 mg decitabine and 100 mg cedazuridine; PO QD)
  Interventions: Drug: Decitabine/cedazuridine

INTERVENTIONS:
Drug: Decitabine/cedazuridine — Decitabine/cedazuridine (INQOVI) oral tablet (35 mg decitabine and 100 mg cedazuridine) taken 3 consecutive days during the first week of every cycle (1 cycle=28-days) for 6 cycles (i.e., 1 course). Additional 6 cycles (i.e., Course 2) for subjects with stable disease or disease regression. Max (total) of 2 treatment courses.

SUMMARY:
This is a Phase II study to determine the rate of stabilization or disease improvement from investigational decitabine/cedazuridine (INQOVI) treatment in subjects with BRCA1-Associated Protein-1 (BAP1) Cancer Predisposition Syndrome (CPDS) and subclinical, early-stage mesothelioma. Progression-free survival (PFS) will also be determined for treated subjects, and the treatment safety (toxicity) evaluated.

DETAILED DESCRIPTION:
Background:

* Mutations involving BRCA1-Associated Protein-1 (BAP1), a nuclear deubiquitinase involved in epigenetic regulation of gene expression, DNA repair, and cellular energetics, have emerged as one of the most common somatic mutations in malignant mesotheliomas.
* Germline mutations involving BAP1 predispose individuals to mesotheliomas and a variety of other malignancies including melanomas, as well as lung, renal, gastric, breast, and hepatobiliary carcinomas.
* The cancer penetrance of germline BAP1 mutations is nearly 100%, and most patients develop multiple synchronous or metachronous neoplasms.
* Mesotheliomas are the most common malignancies diagnosed in subjects with BAP1 Cancer Predisposition Syndrome (CPDS).
* Although clinically evident mesotheliomas arising in the context of germline BAP1 mutations tend to be more indolent than more common, sporadic mesotheliomas, the natural history of early-stage mesotheliomas in subjects with BAP1 CPDS is unknown.
* Presently there are no established guidelines for the treatment of subclinical malignancies in subjects with BAP1 CPDS.
* Epigenetic aberrations including those related to the up regulation of DNA methyltransferases (DNMT) induce genomic instability and enhance the growth and invasion of mesothelioma cells.
* Over-expression of DNMT1 also promotes the development of an immunosuppressive tumor micro-environment (TME).
* Up-regulation of DNMT1 is an early event during mesothelioma development, and levels of DNMT1 over-expression are associated with poor survival in mesothelioma patients.
* Genetic or pharmacologic inhibition of DNMT1 activity induces growth arrest, genomic stress, and apoptosis of mesothelioma cells.
* DNMT1 inhibition can reprogram TMEs thereby promoting more effective antitumor immune responses.
* Decitabine/cedazuridine is an oral DNMT inhibitor which is FDA approved for patients with myelodysplastic syndromes (MDS).
* Conceivably decitabine/cedazuridine therapy can arrest or delay the progression of subclinical/early-stage mesotheliomas in subjects with BAP1 CPDS.

Objective:

-To determine stabilization or disease improvement rates in participants with early-stage mesotheliomas arising in the context of BAP1 CPDS following decitabine/cedazuridine treatment.

Eligibility:

* Participants with history of germline BAP1 mutations and histologically confirmed subclinical, early-stage mesotheliomas, with or without other early-stage BAP1-associated malignancies.
* The extent of the disease insufficient to warrant approved front-line therapies (surgery, chemotherapy, immunotherapy).
* Age >= 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 - 1.
* Willingness to undergo pre- and post-treatment, minimally invasive thoracoscopy, and/or laparoscopy to assess treatment response.
* Adequate cardiac, renal, hepatic, and hematopoietic function.

Design:

* Participants with subclinical, early-stage mesotheliomas will undergo baseline imaging studies followed by minimally invasive thoracoscopy and/or laparoscopy to document the extent of the disease and obtain biopsies for pharmacodynamic (PD) endpoints.
* Participants will then begin oral decitabine/cedazuridine at a fixed dose and schedule (one capsule taken per day for three consecutive days during the first week of each four-week cycle) and will continue this regimen for six cycles.
* Participants will then undergo repeat imaging and minimally invasive thoracoscopy and/or laparoscopy to determine treatment response and obtain tissue for response endpoints.
* Participants who experience disease progression or unacceptable toxicities will be removed from the study.
* Participants with stable disease or disease regression will be offered an additional 6 months of decitabine/cedazuridine treatment.
* Approximately 13 participants will receive study drug on this trial.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Participants with history of germline BRCA1-Associated Protein-1 (BAP1) mutations.
* Histologically confirmed by NCI LP subclinical, early-stage (Tx-T1) mesotheliomas.
* Participants with other early-stage BAP1-associated malignancies in addition to subclinical, early-stage mesotheliomas are eligible for study.
* The extent of the disease (Tx by radiographic imaging) must be insufficient to warrant approved front-line therapies (surgery, chemotherapy, immunotherapy) per standard of care (SOC). Participants with cT1 tumors may be eligible for study if they have been offered and have refused front-line SOC treatment.
* Age >= 18 years.
* Evaluable disease as confirmed by minimally invasive (videoscopic) assessment (thoracoscopy and/or laparoscopy) performed at screening (within 8 weeks prior to treatment initiation).
* Willingness to undergo pre- and post-treatment minimally invasive thoracoscopy and/or laparoscopy to assess treatment response.
* Willingness to co-enroll on 20C0106 (Prospective Evaluation of High Resolution Dual Energy Computed Tomographic Imaging, Noninvasive (Liquid) Biopsies, and Minimally Invasive Surgical Surveillance for Early Detection of Mesotheliomas in Patients with BAP1 Tumor Predisposition Syndrome) and/or 06C0014 (Prospective Evaluation of Genetic and Epigenetic Alterations in Patients with Thoracic Malignancies) to enable collection/processing of tumor, blood and normal pleura if applicable per PI.
* ECOG performance status 0 - 1
* Adequate pulmonary reserve evidenced by FEV1 and DLCO >= 35% predicted on screening pulmonary function testing (PFTs).
* Oxygen saturation >= 92% on room air by pulse oximetry at screening.
* Adequate renal, hepatic, and hematopoietic function at screening as defined below:

  * leukocytes >= 3,000/microL
  * absolute neutrophil count >= 1,500/microL (without transfusion or cytokine support within 2 months prior to study treatment initiation)
  * absolute lymphocyte count > 800/microL
  * platelets >=100,000/microL and < 1,200,000/microL
  * prothrombin time (PT) <=2 seconds above the upper limit of normal (ULN)
  * total bilirubin < 1.5 X institutional upper limit of normal OR direct bilirubin <= 1 ULN for participants with total bilirubin > 1.5 ULN
  * serum albumin >= 2.0 mg/dL
  * aspartate aminotransferase (AST) / alanine aminotransferase (ALT) <= 2.5 X institutional ULN
  * creatinine <= 1.6 mg/ml OR creatinine clearance (eGFR) >= 60 mL/min/1.73 m^2 for participants with creatinine levels above institutional normal.
* Individuals of child-bearing potential (IOCBP) and those that can father children must agree to use an effective method of contraception (barrier, hormonal, intrauterine device (IUD), surgical sterilization) from the study entry and up to 6 months (IOCBP) or 3 months (those that can father children) after the last dose of the decitabine/cedazuridine.
* Nursing (including breastfeeding) participants must be willing to discontinue nursing from study treatment initiation through 2 weeks after the last dose of the study drug.
* The ability of a participant to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* Participants with cancers requiring frontline standard of care treatment.
* Clinically significant cardiovascular/cerebrovascular disease as follows: cerebral vascular accident/stroke (< 6 months prior to study treatment initiation), myocardial infarction (< 6 months prior to study treatment initiation), unstable angina, congestive heart failure (New York Heart Association Classification Class >= II, serious cardiac arrhythmia, clinically significant bleeding or clinically significant pulmonary embolism.
* Therapeutic anticoagulation within 2 weeks prior to study treatment initiation.
* Active Hepatitis A (HAV), Hepatitis B (HBV) (e.g., HBsAg reactive), or Hepatitis C (HCV) (e.g., HCV RNA [qualitative] is detected) at screening.
* History of human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS)-related illness.
* Other active infections requiring systemic therapy.
* Active COVID infection.
* Major surgery within 4 weeks prior to study treatment initiation.
* Immunosuppressive medications within 4 weeks prior to study treatment initiation except non-systemic corticosteroids.
* History of prior treatment with a DNA demethylating agent.
* Pregnancy (confirmed with beta human chorionic gonadotropin (beta-HCG) serum or urine pregnancy test performed in IOCBP at screening).
* Uncontrolled intercurrent illness or situation that would limit compliance with study requirements.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2024-01-31 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
To determine stabilization or disease improvement rates in participants with early-stage mesotheliomas arising in the context of BAP1 CPDS following decitabine/cedazuridine treatment | baseline, before each cycle, after every 6 treatment cycles (Course 1 and Course 2), and at the safety visit
  Assessment of thoracoscopy and/or laparoscopy findings demonstrating stability of evaluable disease or improvement compared to baseline

SECONDARY OUTCOMES:
To evaluate the safety of decitabine/cedazuridine | before each cycle, after every 6 treatment cycles (Course 1 and Course 2), and at the safety visit
  Assessment of safety and tolerability as determined by the frequency and severity of adverse events
To determine PFS in participants receiving decitabine/cedazuridine | baseline, after every 6 treatment cycles (Course 1 and Course 2), and until date of progression or last visit ending at the time of the safety visit
  Progression free survival (PFS) determined by RECIST using the Kaplan-Meier method

CONTACTS AND LOCATIONS:
Overall Officials: David S Schrump, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded will be shared upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data from this study may be requested from other researchers within 10 years after the completion of the primary endpoint by contacting the Principal Investigator.
Access Criteria: Data from this study may be requested by contacting the PI.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_001549-C.html